CLINICAL TRIAL: NCT06362148
Title: Next-Generation Sequencing-based, Tumor- and Plasma-informed Droplet Digital PCR Assay for Detection of Circulating Tumor DNA in Peripheral T-cell Lymphomas
Brief Title: Circulating Tumor DNA in Peripheral T-cell Lymphomas
Acronym: CIRCULATE
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-134-23
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-03

CONDITIONS: Peripheral T-cell Lymphoma; NK/T-Cell Lymphoma
Keywords: Liquid biopsy; Circulating Tumor DNA; ctDNA; Cell Free DNA; cfDNA; mutational profiling
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Extranodal NK-T-Cell | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Diagnostic tumor biopsies Peripheral blood mononuclear cells Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tumor- and plasma-informed, next-generation sequencing (NGS)-based patient-specific droplet digital (dd)PCR assay — Blood sampling for circulating tumor DNA analysis at baseline, cycle 2 day 1, cycle 3 day 1, mid-treatment, end of induction/end of treatment, 100 day follow-up, 6 month, 12 month, 18 month and 24 month follow-up. Blood sampling will also be done in case of relapsing/refractory disease at any point prior to the abovementioned time points.
Diagnostic Test: 18F-fludeoxyglucose positron emission tomography/computed tomography (FDG-PET/CT) — FDG-PET/CT performed at baseline, mid-treatment, end of induction/end of treatment and 6 month, 12 month, 18 month and 24 month follow-up.

SUMMARY:
The aim of this study is to evaluate the feasibility of circulating tumor DNA (ctDNA) measurement in blood plasma for the applicability in prognostication, treatment evaluation and measurable residual disease (MRD) surveillance in a cohort of patients with newly diagnosed or relapsed/refractory peripheral T-cell lymphomas (PTCL).

DETAILED DESCRIPTION:
In this observational prospective cohort study the investigators want to test the use of minimal-invasive liquid biopsies (blood plasma) for the detection of ctDNA in patients with newly diagnosed or relapsed/refractory PTCL. In each enrolled patient a diagnostic tumor-containing tissue biopsy as well as a baseline plasma sample will be subject to targeted next-generation sequencing (NGS) with the aim of identifying tumor-specific genetic alterations and clonal T-cell receptor rearrangements. This testing will be performed on biopsies that have been obtained as a part of standard-of-care diagnostic evaluation for PTCL and no further invasive biopsies will be performed.

Based on the NGS-analysis, a droplet digital polymerase chain reaction (ddPCR) assay will be designed for each patient. ddPCR will be used to detect ctDNA in plasma at diagnosis and later at defined time points during treatment and in the follow-up period.

At the same defined time points PET/CT scans will be performed for later comparative analysis. PTCL patients routinely have PET/CT scans performed before the start of treatment, mid-treatment, at the end of treatment and after hematopoietic stem cell transplant when applicable. PET/CT scans will be conducted every 6 months for the first 2 years of routine follow-up.

Active patient participation (i.e. blood sampling for ctDNA analysis and PET/CT scans) is expected to last up to 27 months from inclusion. Follow-up for survival analysis will be done for up to 5 years from inclusion.

The investigators hypothesize that the NGS-based tumor- and plasma-informed ddPCR assay applied in this study, will provide a highly sensitive and specific tool for prognostication, response evaluation and detection of relapse in patients with PTCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or relapsed/refractory peripheral T-cell lymphoma.
* All primary systemic PTCL entities from the International Consensus Classification 2022.
* ≥18 years of age.
* Life expectancy of 3 months or longer.
* ECOG performance status 0-4 at study entry (PS4 only if lymphoma-induced).
* Measurable disease.
* Written informed consent.

Exclusion Criteria:

* T-cell prolymphocytic leukemia
* T-cell large granular lymphocytic leukemia
* Chronic lymphoproliferative disorder of NK cells
* Adult T-cell leukemia / lymphoma
* Aggressive NK-cell leukemia
* Primary cutaneous T-cell lymphoma such as Sézary syndrome and Mycosis fungoides.
* Primary cutaneous CD30 positive T-cell lymphoproliferative disorders.
* Lymphomatoid papulosis.
* Primary cutaneous anaplastic large cell lymphoma.
* Primary cutaneous small/medium CD4-positive T-cell lymphoproliferative disorder.
* Primary cutaneous gamma-delta T-cell lymphoma.
* Primary cutaneous acral CD8-positive T-cell lymphoproliferative disorder.
* Primary cutaneous CD8-positive aggressive epidermotropic cytotoxic T-cell lymphoma.
* History of active cancer during the past year, except basal cell carcinoma of the skin or stage 0 cervical carcinoma (in situ).
* Unwillingness or inability to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral T-cell lymphomas managed at tertiary care hospitals in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
ctDNA occurrence | Up to 27 months
  Proportion of patients with one or more measurable genetic alterations detected in plasma ctDNA by a tumor-informed, NGS-based patient-specific droplet digital PCR assay at baseline, cycle 2 day 1, cycle 3 day 1, mid-treatment, end of treatment, 6 month, 12 month, 18 month and 24 month follow-up.
ctDNA quantification | Up to 27 months
  Median ctDNA levels in plasma by a tumor- and plasma-informed, NGS-based patient-specific droplet digital PCR assay at baseline, cycle 2 day 1, cycle 3 day 1, mid-treatment, end of treatment, 6 month, 12 month, 18 month and 24 month follow-up.

SECONDARY OUTCOMES:
Progression free survival | Up to 5 years
  Time from date of diagnosis until the date of disease progression or relapse or death from any cause, whichever occurred first.
Overall survival | Up to 5 years
  Time from date of diagnosis to the date of death from any cause or the date of last follow-up. Patients who are event-free at their last follow-up evaluation will be censored at that time point.
Radiographic assessment by PET/CT | Up to 27 months
  Description of tumor staging, metabolic tumor volume and total lesion glycolysis by 18F-fludeoxyglucose positron emission tomography/computed tomography (PET/CT) before treatment. Therapeutic response evaluation based on the 2014 Lugano classification criteria at mid-treatment, end of treatment, 6 month, 12 month, 18 month and 24 month follow-up.
Comparison of molecular and radiographic response | Up to 27 months
  Concordance between detection of ctDNA (MRD-positive or MRD-negative) and therapeutic response assessed by PET/CT at mid-treatment, end of treatment, 6 month, 12 month, 18 month and 24 month follow-up.
Spatial and temporal mutational homo- or heterogeneity | Up to 27 months
  Characterization of the con- or discordance between the genetic profile in tumor and plasma ctDNA at diagnosis and at relapse.
Fragment pattern analysis | Up to 27 months
  Description of fragment sizes of ctDNA by capillary electrophoresis at baseline, cycle 2 day 1, cycle 3 day 1, mid-treatment, end of treatment, 6 month, 12 month, 18 month and 24 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco A d'Amore, MD, DMSc, Study Chair — Aarhus University Hospital and Aarhus University; Patrick R Noerhave, MD, Principal Investigator — Aarhus University Hospital and Aarhus University
Locations (1):
- Department of Hematology, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No